CLINICAL TRIAL: NCT06983288
Title: Perioperative Privacy in the Surgical Patient: A Descriptive Study
Brief Title: Perioperative Privacy in the Surgical Patient
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ezgi Arslan, PhD, Research Assisstant (Principal Investigator), Aydin Adnan Menderes University
Other Study IDs: Perioperative Privacy
Record Dates: First submitted 2025-05-14; First posted 2025-05-21 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Nursing Care; Privacy Statements; Perioperative Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since surgical patients are at risk of privacy violations in the perioperative process, it is thought that determining privacy perceptions and factors affecting this situation and developing strategies to protect privacy will improve the quality of patient care. In this study, it was aimed to determine the privacy perceptions of surgical patients in the perioperative process and the factors affecting them.

DETAILED DESCRIPTION:
Patient privacy is defined as conducting medical procedures and evaluations related to patients' health and disease processes in confidentiality. Patient privacy means not only protecting the information and documents obtained during diagnosis and treatment processes, but also ensuring the confidentiality of the patient's physical body. The most comprehensive regulation on patient privacy in our country is Article 21 of the Patient Rights Regulation, which states that 'it is essential to respect the privacy of the patient, and any medical intervention can be performed by respecting the patient's privacy'. Similarly, the Ministry of Health published a general regulation on 'respecting patient privacy' in 2016, which emphasises that 'it has been observed that patient privacy is not sufficiently respected during examinations, examinations and treatments, especially during surgical procedures and in intensive care units, and the necessary sensitivity should be shown in this regard'. Respecting and protecting the privacy of the patient is one of the basic nursing responsibilities that must be fulfilled during health care delivery.

Both the patient's body privacy and personal information are among the basic nursing values that surgical nurses should protect and implement within the scope of the 'patient advocacy' role. Privacy violations may occur in the preoperative, intraoperative and postoperative processes of patients. In the preoperative period, patients who are admitted to the ward with many symptoms may share the same room with unfamiliar people in unfamiliar rooms, invasive procedures applied to them are performed in a way that they do not want others to see them, identity information and files are shared with more than one person for educational purposes, especially in university hospitals, and the presence of more than one physician or nurse in the room during physical examination may reveal privacy violations. Violations of privacy may also occur for similar reasons during the operation and during the waking process after anaesthesia, such as wearing only underwear during the operation, covering the patient during the operation, not being able to control their own private areas due to the inability to feel part of their body or their whole body due to the effect of anaesthesia.

Patients admitted to hospital for surgery are at risk of privacy violations considering the care practices brought by the surgical process. The possibility of these violations emerges as privacy anxiety in patients. It is thought that it is important to determine the privacy anxiety that occurs in the patient during the surgical process. Although many studies on patient privacy have been conducted in the literature, this study aimed to determine the perioperative privacy levels of patients undergoing surgery in urology, orthopedics, general surgery and gynaecology services.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Knowing and speaking Turkish
* No communication problems
* To have been operated in Aydın Adnan Menderes University Application and Research Hospital Hospital urology, orthopedics, general surgery and gynaecology service
* At least 24 hours since the operation
* To agree to participate in the research

Exclusion Criteria:

* Hospitalisation in the intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Undergoing urology, orthopaedics, general surgery and gynaecology operations
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Privacy perceptions level | Time frame: Postoperative 1st day
  Assessed with Perioperative Privacy Scale. The scale used to evaluate patient perceptions about privacy along perioperative period. It consisted 19 items with scoring from 1 (one) to 5 (five). The maximum score that can be obtained from the scale is 80 and the minimum score is 16. The scale score is high in patients whose privacy is protected and low in patients whose privacy is not protected. The high scores that can be obtained from the scale indicate that the privacy of the patients is protected.

SECONDARY OUTCOMES:
Comfort level | Time frame: Postoperative 1st day
  Assessed with numerical rating scale. The scale used to evaluate patient comfort on postoperative days. The patient were asked to give a score from 1 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Zafer Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 12 months after publication